CLINICAL TRIAL: NCT02766868
Title: Sequential Intensive Chemotherapy With Reduced Intensity Conditioning Regimen in Adult Patients With Refractory and Relapse Acute Lymphoblastic Leukemia
Brief Title: Sequential Intensive Chemotherapy Followed by RIC for Refractory and Relapse ALL
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Principal Investigator, Jiong HU, Head, Blood and Marrow Transplantation Program, Shanghai Jiao Tong University School of Medicine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RJH-2015-RefactoryALL-SCT
Record Dates: First submitted 2016-05-09; First posted 2016-05-10 (Estimated); Last update posted 2016-08-01 (Estimated); Status verified 2016-07

CONDITIONS: Lymphoblastic Leukemia, Acute, Adult
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- FACE-Flu/Bu/Cy (Experimental): Chemotherapy with Fludarabine+cytarabine+cyclophosphamide+etoposie followed by conditioning regimen with Fludarabine, busulfan and Cyclophosphamide
  Interventions: Drug: FACE-Flu/Bu/Cy

INTERVENTIONS:
Drug: FACE-Flu/Bu/Cy — Chemotherapy with Fludarabine+cytarabine+cyclophosphamide+etoposie followed by conditioning regimen with Fludarabine, busulfan and Cyclophosphamide
  Other Names: FACE-chemo-FLu-BU-CY conditioning

SUMMARY:
Patients with refractory and relapse lymphoblastic leukemia had poor outcome even with marrow ablative conditioning mostly standard iv-Bu-Cy or Cy-TBI. In this study, we focus on a new treatment strategy with high-dose chemotherapy regimen consisting of fludaraibine+cytarabine+cyclophosphamide+etoposide followed by reduced intensity condiotning regimen consisting of fludarabine, busulfan and post-infusion cyclophophamide.

DETAILED DESCRIPTION:
All patients with refractory and relapse lymphoblastic leukemia will receive a high-dose chemotherapy regimen consisting of fludaraibine+cytarabine+ cyclophosphamide+etoposide. At day 7 after chemo, a bone marrow aspiration and MRD study by flow-cytometry is planned. For those patients with no residual blasts will undergo allogeneic stem cell transplantation with reduced intensity condiotning regimen consisting of 5-day fludarabine and 3-day busulfan and post-infusion cyclophophamide (D+3 and +4) as GVHD prophylaxis.

ELIGIBILITY:
Inclusion Criteria:

* adult patients with refractory or relapse acute lymphoblastic leukemia not in remission after 2 cycles of induction chemotherapy early relapse (1st remission less than 6 months) not in remission after 1 cycle of re-induction chemotherapy multiple relapse
* age 16-60 years with inform consent
* no contraindication for allogeneic transplantation: active infection, allergy to FLu/Bu/CTX, liver and renal function damage
* HLA matched related (6/6), unrelated donors (8~10/10) or haplo

Exclusion Criteria:

* liver function/renal function damage (over 2 X upper normal range)
* mental disease

Ages: 16 Years to 59 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 20 (Estimated)
Dates: Start 2016-01; Primary Completion 2019-01 (Estimated); Study Completion 2019-07 (Estimated)

PRIMARY OUTCOMES:
disease-free survival | 2 year

CONTACTS AND LOCATIONS:
Overall Officials: Jiong Hu, Principal Investigator — Rui Jin Hospital, Shanghai JiaoTong University School of Medicine
Locations (1):
- Blood & Marrow Transplantation Center, RuiJin Hospital, Shanghai, China

IPD SHARING:
Plan to Share IPD: No